CLINICAL TRIAL: NCT06838221
Title: Interactive Oral Health Educational Program for Children With Intellectual Disability and Their Caregivers.
Acronym: oral program
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Marnal Ahmed Abdelal Elbanna, principal investigator, Cairo University
Other Study IDs: Educational program
Record Dates: First submitted 2025-02-14; First posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Intellectual Disability; Caregiver Burden
Keywords: Interactive oral health educational program
MeSH Terms: conditions — Intellectual Disability; Caregiver Burden | interventions — Lead

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- intellectual disability children and their care givers: oral health educational interactive program of intellectual disabilitry and their care givers
  Interventions: Other: A Before and After study; Other: before and after study

INTERVENTIONS:
Other: A Before and After study — interactive oral health educational program for children with intellectual disability and their care givers
Other: before and after study — To evaluate the oral health of a group of children with disability and determine the effectiveness of the interactive oral health education program on oral health of children and care givers' oral health knowledge.

SUMMARY:
Conducting a research with an interactive oral health educational program and assessing knowledge of caregivers using a questionnaire will help in collecting information about the oral health educational program for children with intellectual disability and the extent of knowledge of care givers in Egypt. This will aid in identifying the knowledge gap, interest, attitude, and practice challenges regarding the children with intellectual disability.

DETAILED DESCRIPTION:
For all children, oral health is a crucial component of overall health, but it is even more crucial for kids with particular medical requirements. Despite the high prevalence of dental disorders among them, people with disabilities or illnesses receive less oral treatment than the general population. According to reports, the largest unmet health need among disabled individuals is dental care. The general health and well-being of the body are closely linked to oral health. The quality of life is enhanced by good dental health. Mentally disabled patients have worse oral health than their normal counterparts, which makes it harder for them to use the oral cavity for activities like eating, swallowing, speaking, chewing, and drooling. This leads to malocclusion, compromised appearance, and poor overall health. Educating parents, guardians, and other caregivers on the causes and self-care prevention of dental disease is a critical part in lowering the caries/gingivitis rate among these children globally. Because of the insufficiency of oral health programs offered in institutions or schools for these particular children, parents and care givers usually have little knowledge about mouth health. they do not understand the significance of dental health, and the educational resources that are accessible to them are frequently insufficient and out-of-date

ELIGIBILITY:
Inclusion Criteria:

* children with intellectual disability
* care givers
* IQ(mild)50-69
* IQ(moderate) 35-49

Exclusion Criteria:

* IQ(severe) 20-34
* refusal to get enrolled in the study.

Ages: 7 Months to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: intellectual disability children and their care givers
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-02-14 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Oral health of children | 3 months
  Oral health of children:
  Gingival index (GL)
  * Before starting the educational program.
  * At the end of the educational program. Score from 0,1,2,3 and Plaque index (PL)
  * Before starting the educational program.
  * At the end of the educational program. Score from 0,1,2,3

SECONDARY OUTCOMES:
Secondary outcome Knowledge of Care givers Questionnaire chart | 3 months
  Secondary outcome Knowledge of Care givers Questionnaire chart
  * Before starting the educational program.
  * At the end of the educational program. Score

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Da'aj, S.T., Al-Bayati, S., Al-Karawi, A.J., & Hameed, A.S. (2023). Oral Health Education (OHE) Program on Adolescents before and after Teacher's Training in Diyala City: A Comparative Clinical Study. The Egyptian Journal of Hospital Medicine.